CLINICAL TRIAL: NCT04017325
Title: A European Randomised Phase 3 Study to Assess the Efficacy and Safety of TOOKAD® Soluble for Localised Prostate Cancer Compared to Active Surveillance. Post Study 5-year Follow-up
Brief Title: European Randomised Study of TOOKAD® Soluble for Prostate Cancer vs Active Surveillance. Post Study Follow-up
Status: Completed | Type: Observational
Sponsor: Steba Biotech S.A. (Other)
Collaborators: International Drug Development Institute (Other); ICON plc (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN1001 PCM301-FU5
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Cancer of the Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TOOKAD VTP TREATMENT: Subjects randomized in the treatment arm (TOOKAD VTP treatment) in the initial period of the study.
  Interventions: Other: no intervention (post study follow up)
- Active surveillance: Subjects randomized in the control group (active surveillance) in the initial period of the study.
  Interventions: Other: no intervention (post study follow up)

INTERVENTIONS:
Other: no intervention (post study follow up) — No intervention (post study follow up)

SUMMARY:
This is an open observational extended follow-up study of patients originally randomized into TOOKAD® Soluble VTP therapy or active surveillance (control group). Additional 60-month follow-up study

DETAILED DESCRIPTION:
This is an open observational extended follow-up study of patients originally randomized into TOOKAD® Soluble VTP therapy or active surveillance (control group). No intervention or further intervention with TOOKAD® Soluble is mandated in this additional 60-month follow-up study where patients in the original TOOKAD® Soluble group and active surveillance (control) group are both managed by their physician as appropriate to their condition using any treatment available following a 'local standard of care' principle from the end of the trial (M24) up to the end of follow-up (M84). Management decisions are entirely left to clinicians and their patients in this pragmatic extension of the trial (no criteria imposed) where standard of care that reflects clinical practice within each centre is applied.

All patients originally randomised in study CLIN1001 PCM301, whether allocated to the TOOKAD® Soluble VTP arm (n=206) or Active surveillance arm (n=207 and who did not withdraw their consent will be included in this extension study.

This extension study consists of 2 different follow-up:

* a follow-up of patients via investigators
* and a follow-up via interviews directly with patients

ELIGIBILITY:
Inclusion Criteria:

* All subjects originally randomized in study CLIN1001 PCM301 are included in this follow-up study. As a reminder, they all met the following criteria at entry (from the original protocol):

  1. Low risk prostate cancer diagnosed using one trans-rectal ultrasound guided biopsy (TRUS) using from 10 to 24 cores, within 12 months of enrolment and showing the following:

     * Gleason 3 + 3 prostate adenocarcinoma as a maximum,
     * Two (2) to three (3) cores positive for cancer. Patients with only one positive core can be included provided they have at least 3 mm of cancer core length.
     * A maximum cancer core length of 5 mm in any core.
  2. Cancer clinical stage up to T2a (pathological or radiological up to T2c disease permitted).
  3. Serum prostate specific antigen (PSA) of 10 ng/mL or less.
  4. Prostate volume equal or greater than 25 cc and less than 70 cc.
  5. Male subjects aged 18 years or older.

Exclusion Criteria:

* As a reminder, all subjects originally randomized did not met the following criteria at entry (from the original protocol):

  1. Unwillingness to accept randomization to either of the two arms of the study.
  2. Any prior or current treatment for prostate cancer, including surgery, radiation therapy (external or brachytherapy) or chemotherapy.
  3. Any surgical intervention for benign prostatic hypertrophy.
  4. Life expectancy less than 10 years.
  5. Any condition or history of illness or surgery that may pose an additional risk to men undergoing the VTP procedure.
  6. Participation in another clinical study or recipient of an investigational product within 1 month of study entry.
  7. Subject unable to understand the patient's information document, to give consent or complete the study tasks. Subject in custody and or in residence in a nursing home or rehabilitation facility.
  8. Contra-indication to MRI (e.g., pacemaker, history of allergic reaction to gadolinium), or factors excluding accurate reading of pelvic MRI (e.g., hip prosthesis).

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients with localized low risk prostate cancer initialy randomized in the study CLIN 1001 PCM301
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Disease progression | Over the 5 years of follow up
  Progression of disease from low risk prostate cancer to moderate or higher risk prostate cancer in men initially randomized to TOOKAD® Soluble VTP compared to men originally randomized on active surveillance.
Other prostate cancer therapy | Over the 5 years of follow up
  Use of other prostate cancer therapy: radical therapy (surgery, radiotherapy, cryotherapy, ultrasound therapy), hormonal therapy or chemotherapy or any therapy indicated for the treatment of prostate cancer in the countries of the study.
Prostate cancer-related death. | Over the 5 years of follow up
  Any death related to Prostate cancer

SECONDARY OUTCOMES:
Absence of cancer | Over the 5 years of follow up
  The proportion of absence of cancer at biopsy (when available)
Radical therapy | Over the 5 years of follow up
  The rate of prostate cancer radical therapy;
Cancer burden | Over the 5 years of follow up
  The total cancer burden in the prostate
Urinary incontinence | Over the 5 years of follow up
  The description of incontinence in terms of mean, median, SD, inter-quartile ranges, min-max
Erectile dysfunction | Over the 5 years of follow up
  The description of erectile dysfunction in terms of mean, median, SD, inter-quartile ranges, min-max
Urethral stenosis | Over the 5 years of follow up
  The rate of urethral stenosis
Prostate cancer complication | Over the 5 years of follow up
  The rate of severe prostate cancer related events: cancer extension to T3, metastasis and prostate cancer related death
Patients Questionnaires Quality of life | Over the 5 years of follow up
  Overal Quality of Life will be recorded for potential utility and descriptives studies

CONTACTS AND LOCATIONS:
Overall Officials: Mark EMBERTON, Professor, Principal Investigator — University College of London Hospital , United Kingdom
Locations (36):
- Department of Urology-Tampere University Hospital-, Tampere, Finland
- France (12):
  - Centre Hospitalier Universitaire (CHU), Angers
  - CHRU Hopital Jean Minjoz, Besançon
  - Site Médipole, Cabestany
  - Polyclinique Sévigné, Cesson-Sévigné
  - Hôpital Claude Huriez, Lille
  - Hôpital La Conception, Marseille
  - Hôpital Tenon, Paris
  - Institut Mutualiste Montsouris (IMM), Paris
  - Hôpital Cochin, Paris
  - Centre Hospitalier Universitaire Lyon Sud, Pierre-Bénite
  - CHU Pontchaillou, Rennes
  - Clinique Urologique Nantes, Saint-Herblain
- Germany (11):
  - Marien Krankenahaus GmbH, Bergisch Gladbach
  - ATURO-Gemeinschaftspraxis für Urologie und Andrologie, Berlin-Wilmersdorf
  - Klinikum Braunschweig, Braunschweig
  - Universitätsklinikum "Carl Gustav Carus" der Technischen Universität, Dresden
  - Urologische Gemeinschaftspraxis, Emmendingen
  - Martini-Klinik am UKE Hamburg-Eppendorf Prostate Cancer Center, Hamburg
  - Vinzenz Krankenhaus - Department of Urology, Hanover
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - University Hospital Schleswig-Holstein, Kiel
  - Ludwig-Maximilians-Universität München, Munich
  - Urologie 24, Nuremberg
- Osp. S. Giov. Battista Molinette-Dipartimento di Discipline Medico-Chirurgiche Urologia, Torino, Italy
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - Catharina Ziekenhuis, Eindhoven
- Spain (4):
  - Hospital Universitario de A Coruña, A Coruña
  - Department of Urology-Hospital Clinic, University of Barcelona, Barcelona
  - Complejo Hospitalario Regional Virgen Del Rocio-Department Urology, Seville
  - Instituto Valenciano de Oncologia, Valencia
- Dept of Urology-University Hospital-, Malmo, Sweden
- United Kingdom (4):
  - Kings College Hospital (KCH), London
  - University College London Hospital (UCLH), London
  - Oxford John Radcliffe Hospital Trust, Oxford
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No